CLINICAL TRIAL: NCT05992298
Title: Explorative Technical Feasibility Testing of 7-Tesla Magnetic Resonance Imaging of the Musculoskeletal System and of the Head
Brief Title: Feasibility Testing of 7-Tesla Magnetic Resonance Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reto Sutter, MD (Other)
Responsible Party: Sponsor-Investigator, Reto Sutter, MD, Prof. Dr. med. Reto Sutter, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I0171
Record Dates: First submitted 2023-07-18; First posted 2023-08-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 7 T MRI (Experimental)
  Interventions: Other: 7 T MRI vs 3 T MRI

INTERVENTIONS:
Other: 7 T MRI vs 3 T MRI — Adult healthy and patient volunteers will undergo a ca. 1 hour examination of non-invasive magnetic-resonance imaging at 7T, and, if appropriate, a closely matching examination at 3T as a standard of reference.

SUMMARY:
The goal of the current project is to explore and develop the technical feasibility of non-invasive imaging of the human musculoskeletal system and head with the first 7T MR scanner with a CE mark to identify areas where the higher field promises significant benefits in qualitative image quality. For a subset of the planned exams, state-of-the art 7T or 3T images will be used as standard of reference to comparatively gauge the qualitative image quality of the investigational 7T images.

ELIGIBILITY:
Inclusion Criteria:

* Consent to undergo a 7T (and, if appropriate a comparative 3T) MRI exam.
* For some of the consistent small series: presence of a specific condition of the musculoskeletal system or of the head. This can include traumatic or degenerative changes, e.g., of tendons, cartilage, muscle, peripheral nerves, ligaments, and bones, or in the brain, as well as focal lesions, e.g., tumors.

Exclusion Criteria:

* Contraindications to undergo a MRI examination at a field strength of 7 Tesla or at 3 Tesla.
* Irregular anatomy and/or tissue properties
* Inability to consent - for any reason.
* Body mass above 200 kg.
* Body mass below 30 kg.
* Women: pregnancy.
* Age below 18.
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Qualitative image quality of 7 T MRI | through study completion, an average of 1 year
  Current-day feasibility of various types of MR examinations of the human musculoskeletal system. The primary outcomes of small consistent series of the study are visual gradings and qualitative measures of image quality. Image quality is rated by independent readers using Likert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Sutter, Prof., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland